CLINICAL TRIAL: NCT03183908
Title: Safety and Immunogenicity of Adjuvanted Versus High-Dose Inactivated Influenza Vaccines in Older Adults
Brief Title: FLUAD® vs. Fluzone® High-Dose Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Boston Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00083845
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Pain; Quality of Life; Injection Site Reaction; Side Effect of Drug; Adverse Drug Event
Keywords: influenza vaccine; fever following vaccination; pain following vaccination; quality of life
MeSH Terms: conditions — Pain; Injection Site Reaction; Drug-Related Side Effects and Adverse Reactions; Influenza, Human | interventions — fluad vaccine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subject, study coordinators, and investigators will be blinded to the type of flu vaccine administered. Only the vaccinator will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Adjuvanted influenza vaccine (FLUAD®) (Active Comparator): In the study arm, subjects will receive a single dose of FLUAD® adjuvanted influenza vaccine during Visit 1.
  Interventions: Biological: FLUAD®
- High-dose influenza vaccine (Fluzone® HD) (Active Comparator): In the study arm, subjects will receive a single dose of Fluzone® High-Dose influenza vaccine during Visit 1.
  Interventions: Biological: Fluzone® High-Dose

INTERVENTIONS:
Biological: FLUAD® — Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
  Other Names: Adjuvanted influenza vaccine
  Arms: Adjuvanted influenza vaccine (FLUAD®)
Biological: Fluzone® High-Dose — Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
  Other Names: High-dose influenza vaccine
  Arms: High-dose influenza vaccine (Fluzone® HD)

SUMMARY:
The overall aim of the study is to compare safety and immunogenicity of inactivated influenza vaccine (IIV), adjuvanted (FLUAD®) versus High-Dose inactivated influenza (Fluzone® High-Dose) vaccine in persons ≥65 years (20% aged ≥80 years). A prospective, randomized, blinded clinical trial that will be conducted during the 2017/2018 and 2018/2019 influenza seasons. During each season, approximately 220 older adults will be enrolled at Duke University Medical Center and 140 older adults at Boston University Medical Center. Eligible subjects will be randomized to receive either adjuvanted influenza vaccine or High-Dose influenza vaccine. All subjects will receive vaccine and provide a blood draw at Visit 1, and then return for a second blood draw without vaccination about 4 weeks later to assess for influenza antibody titers. A subset of 100 subjects at Duke will provide a third blood draw 6 months post-vaccination to assess for waning of influenza antibody titers. Subjects will record the occurrence of local and systemic reactions (including fever, pain, tenderness, swelling, redness, general systemic systems), unsolicited adverse events, medical care utilization, and changes in medications over 8 days following vaccination. In addition, serious adverse events and events of clinical interest will be assessed through 42 days post-vaccination. Health-related quality of life will be assessed pre-vaccination (Day 1) and on Days 3 and 9 post-vaccination.

DETAILED DESCRIPTION:
Full Analysis Population 1: Defined as all subjects who are randomized, vaccinated, and provide at least one day of complete data on the symptom diary.

Full Analysis Population 2: Defined as all subjects who are randomized and vaccinated.

Immunogenicity Population: Defined as subjects who received vaccine, provided baseline and Visit 4 blood draws of acceptable volume and quality within the protocol-defined time frame with no protocol violations affecting immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Persons aged ≥65 years, living in the community
2. Intention of receiving IIV vaccine based on ACIP-CDC guidelines
3. Willing to provide written informed consent prior to initiation of any study procedures
4. Able to speak English
5. Able and willing to complete baseline assessments and questionnaires, and to allow information to be collected from their electronic medical record
6. Able and willing to complete post-vaccine assessments and questionnaires independently or with assistance
7. Able and willing to have blood drawn for the study
8. Able and willing to return in about one month for a follow-up visit including completing questionnaires and having another blood test
9. Access to and ability to use a phone, independently or with assistance
10. Adequate vision and motor skills to complete the diary form independently or with assistance.
11. Not living in a skilled nursing facility/nursing home/long term acute care facility

Exclusion Criteria:

1. IIV receipt during the current influenza season prior to study enrollment
2. Enrolled in this study during the 2017-18 (Year 1) influenza season

   Note: Year 1 study participants will only be enrolled in Year 2 if they are participating in the sub-study on repeat vaccination
3. Has immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 12 months.
4. Has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematologic malignancy*

   *Participants with a history of malignancy may be included if, after previous treatment by surgical excision, chemotherapy or radiation therapy, the participant has been observed for a period that in the investigator's estimation provides a reasonable assurance of sustained cure (not less than 12 months)
5. Thrombocytopenia, bleeding disorder, or anticoagulant use contraindicating intramuscular injection
6. History of febrile illness (> 100.0°F or 37.8°C) within the past 24 hours prior to IIV administration (temporary deferral)
7. Contraindication to IIV receipt including history of severe allergic reaction after a previous dose of any influenza vaccine; or to a vaccine component*, including egg protein; or a latex allergy

   *Formaldehyde, Octylphenol ethoxylate, neomycin, kanamycin, barium, cetyltrimethlyammonium bromide (CTAB)
8. Any history of Guillain-Barré syndrome
9. Mild to severe dementia as determined by the Mini-Cog tool and the Rowland Universal Dementia Assessment Scale (RUDAS)
10. Substance use that could interfere with study compliance
11. Receipt of any inactivated licensed vaccine within 2 weeks, or live attenuated licensed vaccine within 4 weeks prior to enrollment in this study, or planning receipt of any vaccines during the 42-days post-vaccination period (including pneumococcal vaccines)
12. Anyone who is already enrolled or plans to enroll in another clinical trial with an investigational product within 28 days of vaccine receipt. Co-enrollment in observational or behavioral intervention studies are allowed at any time while enrollment in a clinical trial involving an investigational product (other than vaccine) may occur after 30 days following vaccine receipt.
13. Hearing loss determined by the investigators to prevent successful communication over the phone
14. Any condition which, in the opinion of the investigators, may pose a health risk to the subject or interfere with the evaluation of the study objectives.
15. Anyone who is a relative or subordinate of any research study personnel.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 757 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Schmader, MD, Principal Investigator — Duke University; Theresa Harrington, MD, Principal Investigator — Centers for Disease Control and Prevention; Elizabeth Barnett, MD, Principal Investigator — Boston University
Locations (4):
- United States (4):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmader KE, Liu CK, Flannery B, Rountree W, Auerbach H, Barnett ED, Schlaudecker EP, Todd CA, Poniewierski M, Staat MA, Harrington T, Li R, Broder KR, Walter EB. Immunogenicity of adjuvanted versus high-dose inactivated influenza vaccines in older adults: a randomized clinical trial. Immun Ageing. 2023 Jul 1;20(1):30. doi: 10.1186/s12979-023-00355-7. PMID 37393237
- [Derived] Schmader KE, Liu CK, Harrington T, Rountree W, Auerbach H, Walter EB, Barnett ED, Schlaudecker EP, Todd CA, Poniewierski M, Staat MA, Wodi P, Broder KR. Safety, Reactogenicity, and Health-Related Quality of Life After Trivalent Adjuvanted vs Trivalent High-Dose Inactivated Influenza Vaccines in Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jan 4;4(1):e2031266. doi: 10.1001/jamanetworkopen.2020.31266. PMID 33443580

RESULTS

PARTICIPANT FLOW:
Groups:
- Influenza Vaccine, Adjuvanted (FLUAD®): In the study arm, subjects will receive a single dose of FLUAD adjuvanted influenza vaccine during Visit 1.
  FLUAD: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
- High-Dose Influenza Vaccine (Fluzone HD): In the study arm, subjects will receive a single dose of Fluzone High-Dose influenza vaccine during Visit 1.
  Fluzone High-Dose: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
Period: Overall Study
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Started (Full Analysis Population 2) | 378 | 379
Completed (Full Analysis Population 1) | 378 | 377
Not Completed | 0 | 2
Not completed — Missing Symptom Diary Data | 0 | 2

BASELINE CHARACTERISTICS:
Population: The primary analysis population will be the Full Analysis Population 2; defined as all subjects who are randomized and vaccinated.
Groups:
- Adjuvanted Influenza Vaccine (FLUAD): In the study arm, subjects will receive a single dose of FLUAD adjuvanted influenza vaccine during Visit 1.
  FLUAD: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
- Total: Total of all reporting groups
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD) | High-dose Influenza Vaccine (Fluzone HD) | Total
Number analyzed (Participants) | 378 | 379 | 757
Age, Customized [Count of Participants; unit: Participants]
  Age Group: 65-79 Years | 298 | 296 | 594
  Age Group: 80 or More | 80 | 83 | 163
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 207 | 420
  Male | 165 | 172 | 337
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 346 | 351 | 697
  Unknown or Not Reported | 25 | 27 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black only | 70 | 59 | 129
  Race: Other | 22 | 17 | 39
  Race: White Only | 286 | 303 | 589
Region of Enrollment [Number; unit: participants]
  United States | 378 | 379 | 757

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Injection-Site Pain in Arm That Was Vaccinated, Population 1
Description: Comparison of the proportion of subjects reporting moderate/severe injection site pain within the first week post-vaccination in both treatment groups.
Time Frame: Days 1 through 8 post-vaccination
Population: Full Analysis Population 1
Measure: Count of Participants; unit: Participants
Groups:
- Adjuvanted Influenza Vaccine (FLUAD®): In the study arm, subjects will receive a single dose of FLUAD adjuvanted influenza vaccine during Visit 1.
  FLUAD: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
- High-dose Influenza Vaccine (Fluzone® HD): In the study arm, subjects will receive a single dose of Fluzone High-Dose influenza vaccine during Visit 1.
  Fluzone High-Dose: Advisory Committee on Immunization Practices (ACIP) Recommended Vaccine
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 378 | 377
Participants
  None | 297 | 282
  Mild | 69 | 73
  Mod/Severe | 12 | 22
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); The null hypothesis is allV3 is inferior (i.e., allV3 will have higher rates of moderate/severe injection site pain) to IIV3-HD in regards to the proportion of subjects having moderate or severe injection site pain in the first week post vaccination; Test type: Non-Inferiority — The one-sided non-inferiority test with the alpha level set at 0.025 and non-inferiority margin of 5%, stratified by site; Difference in proportions = -2.7, 95% CI 2-sided [-5.8 to 0.4] — The upper bound of a stratified Newcombe binomial confidence interval with Cochran-Mantel-Haenszel weighting of the difference was used

2. Primary Outcome: Number of Participants With Adverse Events of Clinical Interest, Population 2
Description: The frequency and descriptions of adverse events of clinical interest observed in the two treatment groups.
Time Frame: 42 days post-vaccination and compared between the two groups.
Population: Full Analysis Population 2
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 378 | 379
Participants | 0 | 0

3. Primary Outcome: Observed Serious Adverse Events in Both Treatment Groups, Population 2
Description: The frequency and descriptions of serious adverse events observed in the two treatment groups.
  No analytical analysis was completed.
Time Frame: 42 days post-vaccination and compared between the two groups.
Population: Full Analysis Population 2
Measure: Number; unit: SAE Events
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 378 | 379
SAE Events
  Fall | 2 | 0
  Metastatic squamous cell | 0 | 1
  Post-operative ileus | 0 | 1
  Respiratory Failure | 1 | 0
  Stress induced cardiomyopathy | 1 | 0
  TIA | 1 | 0
  Chest Pain | 0 | 1
  Asthma exacerbation | 1 | 0
  Near syncope due to orthostasis | 1 | 0
  Pulmonary emboli | 1 | 0
  Small bowel obstruction | 1 | 0
  SAEs related to study product | 0 | 0
  SAEs not related to study product | 9 | 3
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®); Test type: Other — The comparison of the number of participants with reported SAEs regardless of relationship to study product were made using 95% confidence intervals. Results were reported using exact binomial confidence intervals; Comparison of Frequencies = 2.38, 95% CI 2-sided [1.09 to 4.47]
Statistical Analysis 2: Comparison: High-dose Influenza Vaccine (Fluzone® HD); Test type: Other — [test comment as in outcome 3, analysis 1]; Comparison of Frequencies = .79, 95% CI 2-sided [0.16 to 2.23]

4. Primary Outcome: Number of Participants With H3N2 HAI Seroconversion
Description: H3N2 hemagglutination inhibition assay (HAI) seroconversion: The proportion of subjects achieving H3N2 seroconversion at day 29 (an HAI titer > 1:40 at day 29 if the baseline titer is < 1:10 or a four-fold rise in HAI titer if the baseline titer is > 1:10) in the respective season's vaccine
Time Frame: 29 days post-vaccination
Population: Immunogenicity Population - subjects receiving the study intervention. Participants analyzed include those that provided baseline and Visit 4 blood draws of acceptable volume and quality within the protocol-defined time frame with no protocol violations affecting immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 342 | 338
Participants | 112 | 130
Statistical Analysis 1: Comparison: Influenza Vaccine, Adjuvanted (FLUAD®) vs High-Dose Influenza Vaccine (Fluzone HD); Test type: Non-Inferiority — This objective will be assessed using a one-sided noninferiority test with the alpha level set at 0.025 and noninferiority margin of 10%. The null hypothesis is the allV3 H3N2 seroconversion rate is inferior to IIV3-HD seroconversion rate; p = 0.1245, Cochran-Mantel-Haenszel; Difference in Proportions = -.0579, 97.5% CI 1-sided [lower limit -.1291] — The directional comparison was the lower bound of the confidence interval using a 10% non-inferiority margin

5. Secondary Outcome: Number of Participants With Local Reactions in Arm That Was Vaccinated - Full Study, Population 1
Description: Comparison of local reactions within the first week post-vaccination in both treatment groups.
Time Frame: Days 1 through 8 post-vaccination
Population: Full Analysis Population 1
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 378 | 377
Participants
  Redness: None | 348 | 341
  Redness: Mild | 24 | 23
  Redness: Mod/Severe | 6 | 13
  Shoulder Pain: None | 317 | 326
  Shoulder Pain: Mild | 44 | 36
  Shoulder Pain: Mod/Severe | 17 | 15
  Swelling: None | 335 | 23
  Swelling: Mild | 34 | 26
  Swelling: Mod/Severe | 9 | 328
  Tenderness: None | 201 | 196
  Tenderness: Mild | 150 | 160
  Tenderness: Mod/Severe | 27 | 21
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Redness; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = -1.9, 98% CI 2-sided [-5.0 to 1.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Shoulder Pain; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = 0.5, 98% CI 2-sided [-3.1 to 4.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Swelling; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = -3.7, 98% CI 2-sided [-7.5 to -0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Tenderness; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = 1.6, 98% CI 2-sided [-2.7 to 5.9] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With Local Reactions in Arm That Was Vaccinated - Ages 65 - 79, Population 1
Description: Comparison of local reactions within the first week post-vaccination in both treatment groups by age group.
Time Frame: Days 1 through 8 post-vaccination
Population: Participants 65-79 years of age in Full Analysis Population 1
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 298 | 294
Participants
  Redness: None | 274 | 267
  Redness: Mild | 21 | 17
  Redness: Mod/Severe | 3 | 10
  Shoulder Pain: None | 246 | 249
  Shoulder Pain: Mild | 36 | 33
  Shoulder Pain: Mod/Severe | 16 | 12
  Swelling: None | 264 | 253
  Swelling: Mild | 28 | 22
  Swelling: Mod/Severe | 6 | 19
  Tenderness: None | 157 | 138
  Tenderness: Mild | 117 | 137
  Tenderness: Mod/Severe | 24 | 19
  Injection Site Pain: None | 232 | 210
  Injection Site Pain: Mild | 56 | 65
  Injection Site Pain: Mod/Severe | 10 | 19
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Redness; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -2.4, 95% CI 2-sided [-5.2 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Shoulder Pain; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 1.3, 95% CI 2-sided [-2.3 to 4.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Swelling; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -4.5, 95% CI 2-sided [-8.1 to -1.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Tenderness; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 1.6, 95% CI 2-sided [-2.7 to 5.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Injection Site Pain; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -3.1, 95% CI 2-sided [-6.9 to 0.4] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With Local Reactions in Arm That Was Vaccinated - Ages 80 +, Population 1
Description: Comparison of local reactions within the first week post-vaccination in both treatment groups by age group.
Time Frame: Days 1 through 8 post-vaccination
Population: Participants 80+ years of age in Full Analysis Population 1
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 80 | 83
Participants
  Redness: None | 74 | 74
  Redness: Mild | 3 | 6
  Redness: Mod/Severe | 3 | 3
  Shoulder Pain: None | 71 | 77
  Shoulder Pain: Mild | 8 | 3
  Shoulder Pain: Mod/Severe | 1 | 3
  Swelling: None | 71 | 75
  Swelling: Mild | 6 | 4
  Swelling: Mod/Severe | 3 | 4
  Tenderness: None | 44 | 58
  Tenderness: Mild | 33 | 23
  Tenderness: Mod/Severe | 3 | 2
  Injection Site Pain: None | 65 | 72
  Injection Site Pain: Mild | 13 | 8
  Injection Site Pain: Mod/Severe | 2 | 3
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Redness; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 0.1, 95% CI 2-sided [-7.3 to 7.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Shoulder Pain; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -2.3, 95% CI 2-sided [-9.5 to 5.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Swelling; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -1.2, 95% CI 2-sided [-8.6 to 6.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Tenderness; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 1.4, 95% CI 2-sided [-5.7 to 8.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Injection Site Pain; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -1.2, 95% CI 2-sided [-7.9 to 5.4] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Participants With Systemic Reactions - Full Study Population, Population 1
Description: Comparison of systemic reactions within the first week post-vaccination in both treatment groups.
Time Frame: Days 1 through 8 post-vaccination
Population: Full Analysis Population 1:
  Four missing patient-reported outcome measures for "Fever" outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 378 | 377
Participants
  Arthralgia: None | 340 | 346
  Arthralgia: Mild | 20 | 20
  Arthralgia: Mod/Severe | 18 | 11
  Chills/Shivering: None | 362 | 363
  Chills/Shivering: Mild | 13 | 9
  Chills/Shivering: Mod/Severe | 3 | 5
  Diarrhea: None | 358 | 359
  Diarrhea: Mild | 15 | 9
  Diarrhea: Mod/Severe | 5 | 9
  Fatigue: None | 319 | 337
  Fatigue: Mild | 32 | 25
  Fatigue: Mod/Severe | 27 | 15
  Fever: number analyzed (Participants) | 378 | 373
  Fever: None | 366 | 358
  Fever: Mild | 11 | 12
  Fever: Mod/Severe | 1 | 3
  Headache: None | 335 | 338
  Headache: Mild | 36 | 31
  Headache: Mod/Severe | 7 | 8
  Malaise: None | 332 | 344
  Malaise: Mild | 28 | 22
  Malaise: Mod/Severe | 18 | 11
  Myalgia: None | 334 | 338
  Myalgia: Mild | 25 | 22
  Myalgia: Mod/Severe | 19 | 17
  Nausea: None | 357 | 362
  Nausea: Mild | 19 | 10
  Nausea: Mod/Severe | 2 | 5
  Vomiting: None | 374 | 374
  Vomiting: Mild | 2 | 1
  Vomiting: Mod/Severe | 2 | 2
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Arthralgia; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = 1.8, 98% CI 2-sided [-1.7 to 5.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Chills/Shivering; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = -0.5, 98% CI 2-sided [-2.8 to 2.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Diarrhea; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = -1.1, 98% CI 2-sided [-4.0 to 1.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Fatigue; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = 3.2, 98% CI 2-sided [-0.8 to 7.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Fever; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = 0.5, 98% CI 2-sided [-2.5 to 2.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Headache; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = -0.3, 98% CI 2-sided [-3.0 to 2.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Malaise; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = 1.8, 98% CI 2-sided [-1.7 to 5.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Myalgia; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = 0.5, 98% CI 2-sided [-3.3 to 4.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Nausea; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = -0.8, 98% CI 2-sided [-3.1 to 1.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Vomiting; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.01 level to adjust for multiple comparisons; Difference in proportions = -0.0, 98% CI 2-sided [-1.8 to 1.8] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Number of Participants With System Reactions - Ages 65 - 79, Population 1
Description: Comparison of systemic reactions within the first week post-vaccination in both treatment groups by age group.
Time Frame: Days 1 through 8 post-vaccination
Population: Participants 65-79 years of age in Full Analysis Population 1: Three missing "Fever" outcome values for the Fluzone HD group.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 298 | 294
Participants
  Arthralgia: None | 266 | 266
  Arthralgia: Mild | 16 | 19
  Arthralgia: Mod/Severe | 16 | 9
  Chills/Shivering: None | 283 | 282
  Chills/Shivering: Mild | 12 | 7
  Chills/Shivering: Mod/Severe | 3 | 5
  Diarrhea: None | 280 | 280
  Diarrhea: Mild | 13 | 7
  Diarrhea: Mod/Severe | 5 | 7
  Fatigue: None | 248 | 258
  Fatigue: Mild | 27 | 22
  Fatigue: Mod/Severe | 23 | 14
  Fever: number analyzed (Participants) | 298 | 291
  Fever: None | 288 | 278
  Fever: Mild | 10 | 10
  Fever: Mod/Severe | 0 | 3
  Headache: None | 259 | 257
  Headache: Mild | 32 | 29
  Headache: Mod/Severe | 7 | 8
  Malaise: None | 260 | 264
  Malaise: Mild | 24 | 19
  Malaise: Mod/Severe | 14 | 11
  Myalgia: None | 262 | 261
  Myalgia: Mild | 20 | 19
  Myalgia: Mod/Severe | 16 | 14
  Nausea: None | 280 | 280
  Nausea: Mild | 16 | 9
  Nausea: Mod/Severe | 2 | 5
  Vomiting: None | 294 | 291
  Vomiting: Mild | 2 | 1
  Vomiting: Mod/Severe | 2 | 2
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Arthralgia; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 2.3, 95% CI 2-sided [-1.1 to 5.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Chills/Shivering; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -0.7, 95% CI 2-sided [-3.0 to 2.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Diarrhea; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -0.7, 95% CI 2-sided [-3.5 to 1.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Fatigue; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 2.9, 95% CI 2-sided [-1.1 to 7.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Fever; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -1.0, 95% CI 2-sided [-3.0 to -0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Headache; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -0.4, 95% CI 2-sided [-3.2 to 2.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Malaise; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 0.9, 95% CI 2-sided [-2.5 to 4.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Myalgia; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 0.6, 95% CI 2-sided [-3.1 to 4.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Nausea; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -1.0, 95% CI 2-sided [-3.3 to 1.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Vomiting; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -0.0, 95% CI 2-sided [-1.8 to 1.8] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Number of Participants With System Reactions - Ages 80 +, Population 1
Description: Comparison of systemic reactions within the first week post-vaccination in both treatment groups by age group.
Time Frame: Days 1 through 8 post-vaccination
Population: Participants 80+ years of age in Full Analysis Population 1: One missing "Fever" outcome value in the Fluzone HD group.
  No statistical analysis completed on following Outcomes: Chills/Shivering, Headache, Nausea, Vomiting because none reported in this age group.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 80 | 83
Participants
  Arthralgia: None | 74 | 80
  Arthralgia: Mild | 4 | 1
  Arthralgia: Mod/Severe | 2 | 2
  Chills/Shivering: None | 79 | 81
  Chills/Shivering: Mild | 1 | 2
  Chills/Shivering: Mod/Severe | 0 | 0
  Diarrhea: None | 78 | 79
  Diarrhea: Mild | 2 | 2
  Diarrhea: Mod/Severe | 0 | 2
  Fatigue: None | 71 | 79
  Fatigue: Mild | 5 | 3
  Fatigue: Mod/Severe | 4 | 1
  Fever: number analyzed (Participants) | 80 | 82
  Fever: None | 78 | 80
  Fever: Mild | 1 | 2
  Fever: Mod/Severe | 1 | 0
  Headache: None | 76 | 81
  Headache: Mild | 4 | 2
  Headache: Mod/Severe | 0 | 0
  Malaise: None | 72 | 80
  Malaise: Mild | 4 | 3
  Malaise: Mod/Severe | 4 | 0
  Myalgia: None | 72 | 77
  Myalgia: Mild | 5 | 3
  Myalgia: Mod/Severe | 3 | 3
  Nausea: None | 77 | 82
  Nausea: Mild | 3 | 1
  Nausea: Mod/Severe | 0 | 0
  Vomiting: None | 80 | 83
  Vomiting: Mild | 0 | 0
  Vomiting: Mod/Severe | 0 | 0
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Arthralgia; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 0.05, 95% CI 2-sided [-7.2 to 6.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Diarrhea; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = -2.4, 95% CI 2-sided [-8.1 to -0.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Fatigue; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 3.7, 95% CI 2-sided [-3.6 to 10.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Fever; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 1.2, 95% CI 2-sided [-2.4 to 6.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Malaise; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 5.0, 95% CI 2-sided [2.0 to 12.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Myalgia; Test type: Non-Inferiority — Site-stratified, 5% noninferiority test with a one-sided alpha at the 0.025 level; Difference in proportions = 0.1, 95% CI 2-sided [-7.3 to 7.3] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Quality of Life - Late Life Function & Disability Instrument - Full Population
Description: Change in scores on the Late Life Function & Disability Instrument pre-vaccination to post-vaccination (Day 1 - Day 3) compared between the vaccination groups (Year 1 only). Response choices are ranked 1-5, High Scores indicate better outcomes.
  The Function/Activity Scale measured the amount of difficulty in completing a range of activities, or the amount of help required in doing an activity due to physical or mental heath. : None (5); A little (4) ; Some (3), Quite a lot (2), and Cannot Do (1).
  The Disability/Participation Scale measured participation levels in social, family, and community activities due to physical or mental health. Each question has two parts. For the first part of the question, response choices include: Very often (5), Often (4), Once in a while (3), Almost never (2), Never (1). For the second part of the question, response choices include: Not at all (5), A little (4), Somewhat (3), A lot (2), and Completely (1).
Time Frame: Pre-vaccination (Day 1), 2 days post-vaccination (Day 3)
Population: LLFDI data collected for only one year.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 138 | 141
score on a scale
  Activity Limitation | -1.43 [-2.20 to -0.66] | -2.25 [-2.99 to -1.51]
  Daily Activities | -1.26 [-2.04 to -0.48] | -2.06 [-2.77 to -1.35]
  Basic Mobility | -1.37 [-2.06 to -0.68] | -2.43 [-3.14 to -1.72]
  Participation Restriction | -0.86 [-1.57 to -0.15] | -1.58 [-2.31 to -0.85]
  Social Roles | -0.77 [-1.55 to 0.01] | -1.80 [-2.58 to -1.02]
  Instrumental Roles | -1.08 [-1.82 to -0.34] | -1.66 [-2.41 to -0.91]
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Activity Limitation Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — Non-parametric testing was used to evaluate the changes from baseline to compare between groups. A two-sided alpha level set at 0.01 with no adjustments set for multiple comparisons; p = 0.5862, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Daily Activities Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.5648, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Basic Mobility Changes from Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.4196, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Participation Restriction Changes from Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.2418, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Social Roles Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.0746, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Instrumental Roles Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.5497, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Quality of Life - Late Life Function & Disability Instrument - Ages 65 - 79
Description: as for outcome 11
Time Frame: Pre-vaccination (Day 1), 2 days post-vaccination (Day 3)
Population: Participants 65-79 years of age. LLFDI data collected for only one year.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 119 | 120
score on a scale
  Activity Limitation | -1.35 [-2.20 to -0.50] | -2.12 [-2.91 to -1.33]
  Daily Activities | -1.16 [-2.02 to -0.30] | -1.88 [-2.60 to -1.15]
  Basic Mobility | -1.33 [-2.09 to -.056] | -2.29 [-3.03 to -1.55]
  Participation Restriction | -0.81 [-1.52 to -0.10] | -1.69 [-2.44 to -0.93]
  Social Roles | -0.66 [-1.46 to 0.14] | -1.98 [-2.82 to -1.14]
  Instrumental Roles | -1.00 [-1.74 to -0.27] | -1.70 [-2.47 to -0.93]
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Activity Limitation Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — Non-parametric testing was used to evaluate the changes from baseline to compare between groups. A two-sided alpha level set at 0.05 with no adjustments set for multiple comparisons; p = 0.6278, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Daily Activities Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.5622, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Basic Mobility Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.5538, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Participation Restriction Changes from Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.2310, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Social Roles Changes from Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.0435, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Instrumental Roles Changes from Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.6519, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Quality of Life - Late Life Function & Disability Instrument - Ages 80 +
Description: as for outcome 11
Time Frame: Pre-vaccination (Day 1), 2 days post-vaccination (Day 3)
Population: Participants 80+ years of age. LLFDI data collected for only one year.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 19 | 21
score on a scale
  Activity Limitation | -1.94 [-3.81 to -0.08] | -2.99 [-5.25 to -0.74]
  Daily Activities | -1.86 [-3.74 to 0.03] | -3.13 [-5.65 to -0.61]
  Basic Mobility | -1.62 [-3.22 to -0.02] | -3.23 [-5.58 to -0.88]
  Participation Restriction | -1.17 [-4.00 to 1.67] | -0.97 [-3.54 to 1.60]
  Social Roles | -1.45 [-4.31 to 1.41] | -0.72 [-2.98 to 1.53]
  Instrumental Roles | -1.54 [-4.49 to 1.42] | -1.44 [-4.10 to 1.22]
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Activity Limitation Changes from Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.7483, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Daily Activities Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.7483, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Basic Mobility Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.4953, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Participation Restriction Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.8669, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Social Roles Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.8451, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); Instrumental Roles Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.7376, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Quality of Life - EQ-5D-5L -Full Population
Description: Change in scores on the EuroQOL 5 dimensions-5 level (EQ-5D-5L) pre-vaccination and post-vaccination compared between the vaccination groups (Year 1 only).
  Responses on the EQ-5D-5L measure is converted to a Utility Index that ranges from -0.109 (worst health) to 1.000 (best health).
Time Frame: Pre-vaccination (Day 1), 2 days post-vaccination (Day 3)
Population: EQ-5D-5L data collected for only one year.
Measure: Mean (95% Confidence Interval); unit: Change in score
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 378 | 377
Change in score | -0.054 [-0.064 to -0.044] | -0.053 [-0.063 to -0.044]
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); US Index Score Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.7407, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Quality of Life - EQ-5D-5L - Ages 65 - 79
Description: Change in scores on the EuroQOL 5 dimensions-5 level (EQ-5D-5L) pre-vaccination and post-vaccination compared between the vaccination groups and age group (Year 1 only).
  Responses on the EQ-5D-5L measure is converted to a Utility Index that ranges from -0.109 (worst health) to 1.000 (best health).
Time Frame: Pre-vaccination (Day 1), 2 days post-vaccination (Day 3)
Population: Participants 65-79 years of age. EQ-5D-5L data collected for only one year.
Measure: Mean (95% Confidence Interval); unit: Change in score
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 298 | 296
Change in score | -0.054 [-0.065 to -0.042] | -0.051 [-0.062 to -0.040]
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); US Index Score Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.4032, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Quality of Life - EQ-5D-5L - Ages 80 +
Description: Change in scores on the EuroQOL 5 dimensions-5 level (EQ-5D-5L) pre-vaccination and post-vaccination compared between the vaccination groups and age group (Year 1 only)
  Responses on the EQ-5D-5L measure is converted to a Utility Index that ranges from -0.109 (worst health) to 1.000 (best health).
Time Frame: Pre-vaccination (Day 1), 2 days post-vaccination (Day 3)
Population: Participants 80+ years of age. EQ-5D-5L data collected for only one year.
Measure: Mean (95% Confidence Interval); unit: Change in score
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 80 | 83
Change in score | -0.055 [-0.074 to -0.035] | -0.062 [-0.083 to -0.042]
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); US Index Score Changes from Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.4079, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Quality of Life - EQ VAS -Full Population
Description: Change in scores on the EuroQOL visual analogue scale (EQ VAS) pre-vaccination and post-vaccination compared between the vaccination groups (Year 1 only).
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' (100) and 'the worst health you can imagine' (0).
Time Frame: Pre-vaccination (Day 1), 2 days post-vaccination (Day 3)
Population: EQ VAS data collected for only one year.
Measure: Mean (95% Confidence Interval); unit: Change in score
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 378 | 377
Change in score | -2.222 [-3.379 to -1.065] | -2.496 [-3.452 to -1.539]
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); EQ VAS Changes for Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.7948, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Quality of Life - EQ VAS - Ages 65 - 79
Description: Change in scores on the EuroQOL visual analogue scale (EQ VAS) pre-vaccination and post-vaccination compared between the vaccination groups and age group (Year 1 only).
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' (100) and 'the worst health you can imagine' (0).
Time Frame: Pre-vaccination (Day 1), 2 days post-vaccination (Day 3)
Population: Participants 65-79 years of age.
Measure: Mean (95% Confidence Interval); unit: Change in score
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 298 | 296
Change in score | -2.474 [-3.876 to -1.071] | -2.791 [-3.923 to -1.658]
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); EQ VAS Changes from Day 1 to Day 3 Group Comparisons; Test type: Superiority — Non-parametric testing was used to evaluate the changes from baseline to compare between groups. Alpha level set at 0.05 with no adjustments set for multiple comparisons; p = 0.7953, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Quality of Life - EQ VAS - Ages 80 +
Description: as for outcome 18
Time Frame: Pre-vaccination (Day 1), 2 days post-vaccination (Day 3)
Population: Participants 80+ years of age.
Measure: Mean (95% Confidence Interval); unit: Change in score
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
Number analyzed (Participants) | 80 | 83
Change in score | -1.295 [-2.966 to 0.377] | -1.463 [-3.163 to 0.237]
Statistical Analysis 1: Comparison: Adjuvanted Influenza Vaccine (FLUAD®) vs High-dose Influenza Vaccine (Fluzone® HD); EQ VAS Changes from Day 1 to Day 3 Group Comparisons; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.9329, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Seroconversion - 65 and Older
Description: The proportion of subjects achieving seroconversion at day 29 (an HAI titer > 1:40 at day 29 if the baseline titer is < 1:10 or a four-fold rise in HAI titer if the baseline titer
Time Frame: Day 29 (28 days post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 342 | 338
percentage of participants
  A/H1N1 | 28.1 [23.4 to 33.2] | 26.6 [22.0 to 31.7]
  Influenza B | 18.7 [14.7 to 23.3] | 23.4 [19.0 to 28.3]

21. Secondary Outcome: Seroprotection - 65 and Older
Description: Proportion of subjects with a seroprotective HAI titer (≥ 1:40) pre- and post-immunization at day 29 for each IIV antigen in the respective season's vaccine
Time Frame: Day 29 (28 days post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 342 | 338
percentage of participants
  A/H1N1 - Baseline | 69.6 [64.4 to 74.4] | 66.9 [61.6 to 71.8]
  A/H1N1 - Post-vaccination | 83.3 [79.0 to 87.1] | 83.4 [79.0 to 87.2]
  A/H3N2 - Baseline | 66.7 [61.4 to 71.6] | 65.7 [60.4 to 70.7]
  A/H3N2 - Post-vaccination | 89.8 [86.1 to 92.7] | 88.5 [84.6 to 91.6]
  Influenza B - Baseline | 24.6 [20.1 to 29.5] | 26.9 [22.3 to 32.0]
  Influenza B - Post-vaccination | 44.2 [38.8 to 49.6] | 48.8 [43.4 to 54.3]

22. Secondary Outcome: Geometric Mean HAI Titer - 65 and Older
Description: The geometric mean HAI titer (GMT) for each IIV antigen in the respective season's vaccine
Time Frame: Day 29 (28 days post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: GMT
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 342 | 338
GMT
  A/H1N1 - Baseline | 51.8 [44.5 to 60.3] | 50.8 [43.4 to 59.4]
  A/H1N1 - Post-vaccination | 100.0 [86.6 to 115.6] | 98.0 [84.6 to 113.6]
  A/H3N2 - Baseline | 63.4 [52.8 to 76.1] | 58.5 [48.4 to 70.7]
  A/H3N2 - Post-vaccination | 141.7 [123.2 to 162.9] | 177.3 [152.7 to 205.9]
  Influenza B - Baseline | 13.4 [11.9 to 15.0] | 14.7 [12.9 to 16.7]
  Influenza B - Post-vaccination | 21.6 [18.5 to 25.2] | 27.5 [23.5 to 32.3]

23. Secondary Outcome: Seroconversion - Ages 65-79
Description: The proportion of subjects aged 65-79 achieving seroconversion at day 29 (an HAI titer > 1:40 at day 29 if the baseline titer is < 1:10 or a four-fold rise in HAI titer if the baseline titer
Time Frame: Day 29 (28 days post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 269 | 261
percentage of participants
  A/H1N1 | 29.7 [24.3 to 35.6] | 27.2 [21.9 to 33.0]
  A/H3N2 | 34.2 [28.5 to 40.2] | 39.5 [33.5 to 45.7]
  Influenza B | 19.0 [14.5 to 24.2] | 26.1 [20.8 to 31.8]

24. Secondary Outcome: Seroconversion - Ages 80 and Older
Description: The proportion of subjects ages 80 and older achieving seroconversion at day 29 (an HAI titer > 1:40 at day 29 if the baseline titer is < 1:10 or a four-fold rise in HAI titer if the baseline titer
Time Frame: Day 29 (28 days post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 73 | 77
percentage of participants
  A/H1N1 | 21.9 [13.1 to 33.1] | 24.7 [15.6 to 35.8]
  A/H3N2 | 27.4 [17.6 to 39.1] | 35.1 [24.5 to 46.7]
  Influenza B | 17.8 [9.8 to 28.5] | 14.3 [7.4 to 24.1]

25. Secondary Outcome: Seroprotection - Ages 65-79
Description: Proportion of subjects ages 65-79 with a seroprotective HAI titer (≥ 1:40) pre- and post-immunization at day 29 for each IIV antigen in the respective season's vaccine
Time Frame: Day 29 (28 days post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 269 | 261
percentage of participants
  A/H1N1 - Baseline | 69.9 [64.0 to 75.3] | 65.5 [59.4 to 71.2]
  A/H1N1 - Post-vaccination | 83.6 [78.7 to 87.8] | 82.8 [77.6 to 87.1]
  A/H3N2 - Baseline | 67.3 [61.3 to 72.8] | 65.5 [59.4 to 71.2]
  A/H3N2 - Post-vaccination | 91.4 [87.4 to 94.4] | 88.1 [83.6 to 91.7]
  Influenza B - Baseline | 22.3 [17.5 to 27.8] | 19.9 [15.3 to 25.3]
  Influenza B - Post-vaccination | 42.4 [36.4 to 48.5] | 45.2 [39.1 to 51.5]

26. Secondary Outcome: Seroprotection - Ages 80 and Older
Description: Proportion of subjects ages 80 and older with a seroprotective HAI titer (≥ 1:40) pre- and post-immunization at day 29 for each IIV antigen in the respective season's vaccine
Time Frame: Day 29 (28 days post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 73 | 77
percentage of participants
  A/H1N1 - Baseline | 68.5 [56.6 to 78.7] | 71.4 [60.0 to 81.0]
  A/H1N1 - Post-vaccination | 82.2 [71.5 to 89.9] | 85.7 [75.9 to 92.4]
  A/H3N2 - Baseline | 64.4 [52.3 to 75.1] | 66.2 [54.6 to 76.5]
  A/H3N2 - Post-vaccination | 83.6 [73.0 to 91.0] | 89.6 [80.6 to 95.2]
  Influenza B - Baseline | 32.9 [22.3 to 44.8] | 50.6 [39.0 to 62.2]
  Influenza B - Post-vaccination | 50.7 [38.7 to 62.5] | 61.0 [49.2 to 71.8]

27. Secondary Outcome: Geometric Mean HAI Titer - Ages 65-79
Description: The geometric mean HAI titer (GMT) for each IIV antigen in the respective season's vaccine for ages 65-79
Time Frame: Day 29 (28 days post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: GMT
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 269 | 261
GMT
  A/H1N1 - Baseline | 52.5 [44.3 to 62.2] | 49.5 [41.4 to 59.0]
  A/H1N1 - Post-vaccination | 108.8 [92.1 to 128.5] | 100.9 [84.9 to 119.9]
  A/H3N2 - Baseline | 63.3 [51.7 to 77.5] | 56.4 [45.5 to 69.8]
  A/H3N2 - Post-vaccination | 145.3 [124.3 to 169.7] | 184.4 [155.2 to 219.1]
  Influenza B - Baseline | 12.2 [10.8 to 13.8] | 11.8 [10.3 to 13.4]
  Influenza B - Post-vaccination | 20.3 [17.2 to 24.1] | 23.8 [20.0 to 28.4]

28. Secondary Outcome: Geometric Mean HAI Titer - Ages 80 and Older
Description: The geometric mean HAI titer (GMT) for each IIV antigen in the respective season's vaccine for ages 80 and older
Time Frame: Day 29 (28 days post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: GMT
Arm/Group | Influenza Vaccine, Adjuvanted (FLUAD®) | High-Dose Influenza Vaccine (Fluzone HD)
Number analyzed (Participants) | 73 | 77
GMT
  A/H1N1 - Baseline | 49.3 [35.1 to 69.3] | 55.6 [39.2 to 78.8]
  A/H1N1 - Post-vaccination | 73.4 [55.2 to 97.7] | 88.7 [66.7 to 118.0]
  A/H3N2 - Baseline | 63.7 [41.4 to 98.0] | 66.5 [43.9 to 101.0]
  A/H3N2 - Post-vaccination | 129.2 [93.4 to 178.8] | 155.0 [114.2 to 210.5]
  Influenza B - Baseline | 18.7 [14.6 to 24.0] | 31.2 [23.2 to 42.1]
  Influenza B - Post-vaccination | 27.0 [19.0 to 38.2] | 45.0 [31.8 to 63.5]

ADVERSE EVENTS:
Time Frame: Adverse Events, Serious Adverse Events, and All-Cause Mortality rates were collected 42 days post vaccination. Serious Adverse Events and Mortality Rates were collected up to 181 days for the longer-term immunogenicity subset
Description: The two reported deaths occurred >42 days post vaccination
Arm/Group | Adjuvanted Influenza Vaccine (FLUAD®) | High-dose Influenza Vaccine (Fluzone® HD)
All-Cause Mortality (participants affected / at risk) | 1/378 | 1/379
Serious Adverse Events (participants affected / at risk) | 10/378 | 4/379
Other Adverse Events (participants affected / at risk) | 15/378 | 19/379
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvanted Influenza Vaccine (FLUAD®) (N=378) | High-dose Influenza Vaccine (Fluzone® HD) (N=379)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1)
Fall (General disorders) | 2 (2) | 0 (0)
Metastatic squamous cell (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Post-operative ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stressed induced cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
TIA (Nervous system disorders) | 1 (1) | 0 (0)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Near syncope due to orthostatic (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvanted Influenza Vaccine (FLUAD®) (N=378) | High-dose Influenza Vaccine (Fluzone® HD) (N=379)
Cold (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 19 (19) — Cold symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT03183908/Prot_SAP_000.pdf